CLINICAL TRIAL: NCT02260557
Title: A Multi-center, Double-blind, Randomized, Placebo-controlled, Parallel Group, Exploratory Phase 2 Study to Assess Efficacy and Safety of Selexipag in Adult Subjects With Raynaud's Phenomenon Secondary to Systemic Sclerosis
Brief Title: Effects of Selexipag in Adults With Raynaud's Phenomenon Secondary to Systemic Sclerosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Actelion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AC-065C202
Record Dates: First submitted 2014-10-06; First posted 2014-10-09 (Estimated); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Raynaud's Phenomenon Secondary to Systemic Sclerosis
Keywords: Systemic Sclerosis; Raynaud's Phenomenon
MeSH Terms: conditions — Scleroderma, Systemic; Raynaud Disease | interventions — selexipag

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Selexipag (Experimental): Selexipag is initiated at 200 µg twice daily (b.i.d.) and up-titrated every 3 days in 200 μg b.i.d. increments up to the maximum tolerated dose (MTD) for each individual patient but not above 1600 µg during the 3-week titration phase. This is followed by a 5-week maintenance phase, during which patients continue the treatment at their individual MTD.
  Interventions: Drug: Selexipag
- Placebo (Experimental): Placebo matching selexipag tablets is administered according to the same schedule as selexipag
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Selexipag — Film-coated tablets containing 200 μg of selexipag to be administered orally twice daily
  Other Names: ACT-293987
  Arms: Selexipag
Drug: Placebo — Placebo matching selexipag 200 μg tablets to be administered orally twice daily
  Arms: Placebo

SUMMARY:
The primary objective of the study is to determine the activity of selexipag on Raynaud attack frequency in subjects with Raynaud's Phenomenon (RP) secondary to Systemic Sclerosis (SSc).

ELIGIBILITY:
Key inclusion criteria:

* Signed informed consent prior to any study-mandated procedure.
* Male and female subjects aged 18 years and above with a history of recurrent multiple weekly RP attacks secondary to SSc.
* Women of childbearing potential must agree to use a reliable method of birth control.

Key exclusion criteria:

* Known moderate or severe hepatic impairment (i.e. Child-Pugh C).
* Known hypersensitivity to selexipag or drugs of the same class, or any of their excipients.
* Subjects who have received prostacyclin (epoprostenol) or prostacyclin analogs (i.e., treprostenol, iloprost, beraprost) within 3 months prior to the screening visit.
* Subjects who have received a Phosphodiesterase type 5 (PDE-5) inhibitor within 1 week prior to the screening visit.
* Any dose change or initiation of any of the following drugs within 1 month prior to the screening visit: Calcium channel blockers, Nitrates or nitric oxide donors, ERA's, Alpha-blockers, Antithrombotic agents, NSAIDs (occasional use allowed), Angiotensin Converting Enzyme (ACE) inhibitors, Beta-blockers, Clonidine, Systemic corticosteroids, Fluoxetine.
* Severe renal insufficiency (at randomization).
* Any circumstances or conditions, which, in the opinion of the investigator, may affect the subject's full participation in the study or compliance with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2014-10; Primary Completion 2015-04 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Average number of Raynaud's phenomenon (RP) attacks per week during the maintenance treatment period | From Day 26 to Day 56 ( +/- 7 days)
  The number of RP attacks is determined from daily entries in electronic Diaries (eDiary).

SECONDARY OUTCOMES:
Number of patients with treatment-emergent adverse events | Up to end of study (Day 86 +/- 7 days)
  A treatment-emergent adverse event is any adverse event (AE) temporally associated with the use of a study treatment, whether or not considered related to the study treatment, including any abnormalities in ECG parameters, vital signs or laboratory tests
Number of patients with treatment-emergent serious adverse events | Up to end of study (Day 86 +/- 7 days)

OTHER OUTCOMES:
Change from baseline in quality of life (QOL) | At baseline (Day 1) and end of treatment (Day 56 +/- 7 days)
  QOL is assessed by the Scleroderma Health Assessment Questionnaire (SHAQ)

CONTACTS AND LOCATIONS:
Overall Officials: Ralph Preiss, MD, Study Chair — Actelion

REFERENCES:
- [Derived] Denton CP, Hachulla E, Riemekasten G, Schwarting A, Frenoux JM, Frey A, Le Brun FO, Herrick AL; Raynaud Study Investigators. Efficacy and Safety of Selexipag in Adults With Raynaud's Phenomenon Secondary to Systemic Sclerosis: A Randomized, Placebo-Controlled, Phase II Study. Arthritis Rheumatol. 2017 Dec;69(12):2370-2379. doi: 10.1002/art.40242. PMID 29193819